CLINICAL TRIAL: NCT03889639
Title: A Phase 2b Dose-finding Study for SAR442168, a Bruton's Tyrosine Kinase Inhibitor, in Participants With Relapsing Multiple Sclerosis
Brief Title: Dose-finding Study for SAR442168 in Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DRI15928; 2018-003927-12 (EudraCT Number); U1111-1220-0572 (Other: UTN)
Record Dates: First submitted 2019-03-01; First posted 2019-03-26 (Actual); Results first posted 2023-03-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Relapsing Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: SAR442168 5 mg Then Placebo (Experimental): Participants received SAR442168 5 milligrams (mg), orally once daily for first 12 weeks then crossed over to matching placebo orally once daily for 4 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 1: SAR442168 15 mg Then Placebo (Experimental): Participants received SAR442168 15 mg, orally once daily for first 12 weeks then crossed over to matching placebo orally once daily for 4 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 1: SAR442168 30 mg Then Placebo (Experimental): Participants received SAR442168 30 mg, orally once daily for first 12 weeks then crossed over to matching placebo orally once daily for 4 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 1: SAR442168 60 mg Then Placebo (Experimental): Participants received SAR442168 60 mg, orally once daily for first 12 weeks then crossed over to matching placebo orally once daily for 4 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 2: Placebo Then SAR442168 5 mg (Experimental): Participants received placebo matching to SAR442168 tablets, orally once daily for first 4 weeks then crossed over to SAR442168 5 mg orally once daily for 12 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 2: Placebo Then SAR442168 15 mg (Experimental): Participants received placebo matching to SAR442168 tablets, orally once daily for first 4 weeks then crossed over to SAR442168 15 mg orally once daily for 12 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 2: Placebo Then SAR442168 30 mg (Experimental): Participants received placebo matching to SAR442168 tablets, orally once daily for first 4 weeks then crossed over to SAR442168 30 mg orally once daily for 12 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)
- Cohort 2: Placebo Then SAR442168 60 mg (Experimental): Participants received placebo matching to SAR442168 tablets, orally once daily for first 4 weeks then crossed over to SAR442168 60 mg orally once daily for 12 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
  Interventions: Drug: SAR442168; Drug: Placebo; Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI)

INTERVENTIONS:
Drug: SAR442168 — Pharmaceutical form: Film coated tablet; Route of administration: Oral
Drug: Placebo — Pharmaceutical form: Film coated tablet; Route of administration: Oral
Drug: Locally approved intravenous contrast medium for contrast enhanced magnetic resonance imaging (MRI) — Pharmaceutical form: Solution for injection; Route of administration: Intravenous

SUMMARY:
Primary Objective:

To determine the dose-response relationship for SAR442168 to reduce the number of new active brain lesions.

Secondary Objectives:

* To evaluate efficacy of SAR442168 on disease activity as assessed by imaging measures.
* To evaluate the safety and tolerability of SAR442168.

DETAILED DESCRIPTION:
The total study duration was 24 weeks which included a screening period of 4 weeks, a treatment period of 16 weeks, and a follow-up period of up to 4 weeks. Participants who completed the Week 16 visit were proposed to be enrolled in a long-term extension safety and efficacy study to assess safety, tolerability and efficacy of SAR442168.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 55 years of age, inclusive, at the time of signing the informed consent.
* Participant was diagnosed with relapsing multiple sclerosis (RMS) according to the 2017 revision of the McDonald diagnostic criteria.
* Participant must had at least 1 documented relapse within the previous year, OR greater than or equal to (>=) 2 documented relapses within the previous 2 years, OR >=1 active Gadolinium (Gd) enhancing brain lesion on an MRI scan in the past 6 months and prior to screening.
* A female participant must had used a double contraception method including a highly effective method of birth control from inclusion and up to 2 months after the last study dose, except if she had undergone sterilization at least 3 months earlier or was postmenopausal. Menopause was defined as being amenorrheic for >=12 months with serum follicle-stimulating hormone (FSH) level greater than (>) 30 International Units per liters.
* Male participants, whose partners were of childbearing potential (including breastfeeding women), must had accepted to use, during sexual intercourse, a double contraceptive method according to the following algorithm: (condom) plus (intrauterine device or hormonal contraceptive) from inclusion up to 3 months after the last dose.
* Male participants whose partners were pregnant must had used, during sexual intercourse, a condom from inclusion up to 3 months after the last dose.
* Male participants had agreed not to donate sperm from the inclusion up to 3 months after the last dose.
* Participant had given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria:

* The participant had been diagnosed with primary progressive multiple sclerosis according to the 2017 revision of the McDonald diagnostic criteria or with non relapsing secondary progressive multiple sclerosis.
* Requirement for concomitant treatment that could bias the primary evaluation.
* Contraindication for MRI.
* Contraindications to use MRI Gd contrast-enhancing preparations.
* History of infection with the human immunodeficiency virus (HIV).
* History of active or latent tuberculosis.
* Any other active infections that would adversely affect participation or investigational medicinal product administration in this study, as judged by the Investigator.
* Presence of any screening laboratory or electrocardiogram values outside normal limits that were considered in the Investigator's judgment to be clinically significant.
* Presence of liver injury.
* At screening, the participant was positive for hepatitis B surface antigen and/or hepatitis B core antibody and/or was positive for hepatitis C antibody.
* Bleeding disorder or known platelet dysfunction at any time prior to screening visit.
* Participant had received any live (attenuated) vaccine (including but not limited to varicella zoster, oral polio, and nasal influenza) within 2 months before first treatment visit.
* Participant was receiving strong inducers or inhibitors of cytochrome P450 3A (CYP3A) or CYP2C8 hepatic enzymes.
* Participant was receiving anticoagulant/antiplatelet therapies.
* Participant had taken other investigational drugs within 3 months or 5 half lives, whichever was longer, before screening visit.
* Participant had an Expanded Disability Status Scale score >5.5 at first screening visit.
* Participant had a relapse in the 30 days prior to randomization.
* Participant was pregnant or a breastfeeding woman.
* History or presence of significant other concomitant illness.
* The participant had received medications/treatments for multiple sclerosis within a specified time frame.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (48):
- United States (9):
  - Investigational Site Number 8400005, Cullman, Alabama
  - Investigational Site Number 8400002, Maitland, Florida
  - Investigational Site Number 8400004, Sunrise, Florida
  - Investigational Site Number 8400009, Tampa, Florida
  - Investigational Site Number 8400007, Savannah, Georgia
  - Investigational Site Number 8400001, Northbrook, Illinois
  - Investigational Site Number 8400008, Dayton, Ohio
  - Investigational Site Number 8400006, Westerville, Ohio
  - Investigational Site Number 8400003, Knoxville, Tennessee
- Canada (3):
  - Investigational Site Number 1240002, Gatineau
  - Investigational Site Number 1240001, Greenfield Park
  - Investigational Site Number 1240003, Vancouver
- Czechia (7):
  - Investigational Site Number 2030007, Brno
  - Investigational Site Number 2030004, Hradec Králové
  - Investigational Site Number 2030003, Jihlava
  - Investigational Site Number 2030005, Ostrava - Poruba
  - Investigational Site Number 2030006, Pardubice
  - Investigational Site Number 2030001, Prague
  - Investigational Site Number 2030002, Praha 5 - Motol
- Investigational Site Number 2330001, Tallinn, Estonia
- France (4):
  - Investigational Site Number 2500004, Nancy
  - Investigational Site Number 2500001, Nantes
  - Investigational Site Number 2500002, Strasbourg
  - Investigational Site Number 2500003, Toulouse
- Netherlands (2):
  - Investigational Site Number 5280001, Amsterdam
  - Investigational Site Number 5280002, Sittard-Geleen
- Russia (7):
  - Investigational Site Number 6430006, Kazan'
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430005, Saint Petersburg
  - Investigational Site Number 6430004, Saint Petersburg
  - Investigational Site Number 6430001, Saint Petersburg
  - Investigational Site Number 6430007, Tyumen
- Slovakia (2):
  - Investigational Site Number 7030001, Bratislava
  - Investigational Site Number 7030002, Martin
- Spain (6):
  - Investigational Site Number 7240006, Barakaldo
  - Investigational Site Number 7240002, Barcelona
  - Investigational Site Number 7240001, Madrid
  - Investigational Site Number 7240004, Murcia
  - Investigational Site Number 7240005, Salt
  - Investigational Site Number 7240003, Seville
- Ukraine (7):
  - Investigational Site Number 8040002, Chernivtsi
  - Investigational Site Number 8040005, Dnipro
  - Investigational Site Number 8040001, Lviv
  - Investigational Site Number 8040006, Lviv
  - Investigational Site Number 8040009, Odesa
  - Investigational Site Number 8040003, Vinnytsia
  - Investigational Site Number 8040007, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Reich DS, Arnold DL, Vermersch P, Bar-Or A, Fox RJ, Matta A, Turner T, Wallstrom E, Zhang X, Mares M, Khabirov FA, Traboulsee A; Tolebrutinib Phase 2b Study Group. Safety and efficacy of tolebrutinib, an oral brain-penetrant BTK inhibitor, in relapsing multiple sclerosis: a phase 2b, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2021 Sep;20(9):729-738. doi: 10.1016/S1474-4422(21)00237-4. PMID 34418400
- See also: DRI15928 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25224&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 44 active centers in 10 countries. A total of 168 participants were screened from 29-March-2019 to 29-August-2019, of which 38 participants were screen failures. Screen failures were mainly due to selection criteria not met.
Pre-assignment Details: A total of 130 participants were randomized and treated in this study. Participants were centrally assigned to 1 of 8 arms (4 dose groups at an equal ratio to start with SAR442168 [all considered as Cohort 1] or placebo [all considered as Cohort 2]).
Period: Overall Study
Arm/Group | Cohort 1: SAR442168 5 mg Then Placebo | Cohort 1: SAR442168 15 mg Then Placebo | Cohort 1: SAR442168 30 mg Then Placebo | Cohort 1: SAR442168 60 mg Then Placebo | Cohort 2: Placebo Then SAR442168 5 mg | Cohort 2: Placebo Then SAR442168 15 mg | Cohort 2: Placebo Then SAR442168 30 mg | Cohort 2: Placebo Then SAR442168 60 mg
Started | 16 | 16 | 16 | 16 | 17 | 16 | 17 | 16
Completed | 16 | 16 | 16 | 16 | 17 | 16 | 17 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on randomized population that included any participant who had been allocated to a randomly assigned treatment, regardless of whether the treatment kit was used.
Groups:
- Cohort 1: SAR442168 5 mg Then Placebo: Participants received SAR442168 5 mg, orally once daily for first 12 weeks then crossed over to matching placebo orally once daily for 4 weeks during the 16 weeks treatment period. To maintain the blinding, each participant was given a total of 4 tablets daily, either of SAR442168 or SAR442168 and placebo, to achieve the specified daily dose of SAR442168.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SAR442168 5 mg Then Placebo | Cohort 1: SAR442168 15 mg Then Placebo | Cohort 1: SAR442168 30 mg Then Placebo | Cohort 1: SAR442168 60 mg Then Placebo | Cohort 2: Placebo Then SAR442168 5 mg | Cohort 2: Placebo Then SAR442168 15 mg | Cohort 2: Placebo Then SAR442168 30 mg | Cohort 2: Placebo Then SAR442168 60 mg | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 17 | 16 | 17 | 16 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (11.1) | 35.1 (7.9) | 40.8 (8.7) | 38.1 (9.1) | 34.8 (8.6) | 36.7 (10.7) | 37.5 (11.6) | 36.1 (8.7) | 37.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 11 | 15 | 16 | 11 | 10 | 9 | 91
  Male | 7 | 6 | 5 | 1 | 1 | 5 | 7 | 7 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 6
  White | 15 | 15 | 13 | 15 | 17 | 14 | 16 | 14 | 119
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Brain Magnetic Resonance Imaging (MRI) Assessment: Number of New Gadolinium (Gd) Enhancing T1-hyperintense Lesions
Description: Number of new Gd-enhancing T1-hyperintense lesions was detected by brain MRI at the end of 12 weeks of SAR442168 treatment (i.e., at Week 12 for Cohort 1 participants and Week 16 for Cohort 2 participants). Data was planned to be collected and analyzed on pooled population of participants at each dose level of SAR442168 (either in Cohort 1 and 2) and pooled population of participants receiving placebo in Cohort 2 and was not planned to collected during placebo administration in Cohort 1 (Weeks 12 to 16).
Time Frame: After 12 weeks of SAR442168 treatment for SAR442168 reporting arms (i.e., at Week 12 for Cohort 1 participants, at Week 16 for Cohort 2 participants) and at Week 4 for Cohort 2 placebo
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all randomly assigned participants exposed to the study drug, analyzed according to the treatment assigned by randomization. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Cohort 2: Pooled Placebo: All participants in Cohort 2 who received placebo matching to SAR442168 orally once daily for first 4 weeks during the 16 weeks treatment period.
- Cohorts 1 and 2: SAR442168 5 mg: All participants who received SAR442168 5 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohorts 1 and 2: SAR442168 15 mg: All participants who received SAR442168 15 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohorts 1 and 2: SAR442168 30 mg: All participants who received SAR442168 30 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohorts 1 and 2: SAR442168 60 mg: All participants who received SAR442168 60 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
Arm/Group | Cohort 2: Pooled Placebo | Cohorts 1 and 2: SAR442168 5 mg | Cohorts 1 and 2: SAR442168 15 mg | Cohorts 1 and 2: SAR442168 30 mg | Cohorts 1 and 2: SAR442168 60 mg
Number analyzed (Participants) | 59 | 31 | 31 | 33 | 31
lesions | 1.03 (2.50) | 1.39 (3.20) | 0.77 (1.48) | 0.76 (3.31) | 0.13 (0.43)
Statistical Analysis 1: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 5 mg; SAR442168 5 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 5 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95 percentage (%) confidence interval (CI) were reported. Analysis was performed using a negative binomial regression model adjusted for Baseline gadolinium-enhancing T1-hyperintense lesion activity (presence/absence); p = 0.1673, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = -56.16, 95% CI 2-sided [-193.99 to 17.05]
Statistical Analysis 2: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 15 mg; SAR442168 15 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 15 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model adjusted for Baseline gadolinium-enhancing T1-hyperintense lesion activity (presence/absence); p = 0.3540, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = -62.80, 95% CI 2-sided [-356.24 to 41.91]
Statistical Analysis 3: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 30 mg; SAR442168 30 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 30 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model adjusted for Baseline gadolinium-enhancing T1-hyperintense lesion activity (presence/absence); p = 0.7674, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 13.49, 95% CI 2-sided [-126.05 to 66.89]
Statistical Analysis 4: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 60 mg; SAR442168 60 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 60 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model adjusted for Baseline gadolinium-enhancing T1-hyperintense lesion activity (presence/absence); p = 0.0178, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 85.02, 95% CI 2-sided [28.02 to 96.88]

2. Secondary Outcome: Number of New or Enlarging T2 Lesions
Description: Number of new and enlarging T2 lesions was detected by brain MRI at the end of 12 weeks of SAR442168 treatment (i.e., at Week 12 for Cohort 1 participants and Week 16 for Cohort 2 participants).
Time Frame: After 12 weeks of SAR442168 treatment for SAR442168 reporting arms (i.e., at Week 12 for Cohort 1 participants, at Week 16 for Cohort 2 participants), and at Week 4 for Cohort 2 placebo
Population: Analysis was performed on mITT population. Data was planned to be collected and analyzed on pooled population of participants at each dose level of SAR442168 (either in Cohort 1 and 2) and pooled population of participants receiving placebo in Cohort 2 and was not planned to be collected during placebo administration in Cohort 1 (Week 12 to 16). Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cohort 2: Pooled Placebo | Cohorts 1 and 2: SAR442168 5 mg | Cohorts 1 and 2: SAR442168 15 mg | Cohorts 1 and 2: SAR442168 30 mg | Cohorts 1 and 2: SAR442168 60 mg
Number analyzed (Participants) | 59 | 31 | 31 | 33 | 31
lesions | 2.12 (5.16) | 1.90 (3.97) | 1.32 (1.83) | 1.30 (4.90) | 0.23 (0.62)
Statistical Analysis 1: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 5 mg; SAR442168 5 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 5 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model without adjusting for Baseline T2 lesion activity as all participants had at least one T2 lesion at Baseline; p = 0.7736, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 10.17, 95% CI 2-sided [-86.49 to 56.73]
Statistical Analysis 2: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 15 mg; SAR442168 15 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 15 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model without adjusting for Baseline T2 lesion activity as all participants had at least one T2 lesion at Baseline; p = 0.2480, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 37.07, 95% CI 2-sided [-38.08 to 71.32]
Statistical Analysis 3: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 30 mg; SAR442168 30 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 30 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model without adjusting for Baseline T2 lesion activity as all participants had at least one T2 lesion at Baseline; p = 0.3081, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 38.5, 95% CI 2-sided [-56.61 to 75.85]
Statistical Analysis 4: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 60 mg; SAR442168 60 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 60 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model without adjusting for Baseline T2 lesion activity as all participants had at least one T2 lesion at Baseline; p = 0.0001, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 89.34, 95% CI 2-sided [68.39 to 96.41]

3. Secondary Outcome: Total Number of Gd-enhancing T1-hyperintense Lesions
Description: Total number of Gd-enhancing T1-hyperintense lesions was detected by brain MRI at the end of 12 weeks of SAR442168 treatment (i.e., at Week 12 for Cohort 1 participants and Week 16 for Cohort 2 participants).
Time Frame: as for outcome 2
Population: Analysis was performed on mITT population. Data was planned to be collected and analyzed on pooled population of participants at each dose level of SAR442168 (either in Cohort 1 and 2) and pooled population of participants receiving placebo in Cohort 2 and was not planned to be collected during placebo administration in Cohort 1 (Weeks 12 to 16). Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cohort 2: Pooled Placebo | Cohorts 1 and 2: SAR442168 5 mg | Cohorts 1 and 2: SAR442168 15 mg | Cohorts 1 and 2: SAR442168 30 mg | Cohorts 1 and 2: SAR442168 60 mg
Number analyzed (Participants) | 59 | 31 | 31 | 33 | 31
lesions | 1.36 (3.52) | 1.77 (4.10) | 0.87 (1.59) | 1.18 (4.87) | 0.29 (0.86)
Statistical Analysis 1: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 5 mg; SAR442168 5 mg/Placebo; Test type: Superiority — Relative reduction in lesions in SAR442168 5 mg (Cohorts 1 and 2) when compared with placebo (Cohort 2) with 95% CI were reported. Analysis was performed using a negative binomial regression model adjusted for Baseline gadolinium-enhancing T1-hyperintense lesion activity (presence/absence); p = 0.1525, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = -62.16, 95% CI 2-sided [-214.44 to 16.38]
Statistical Analysis 2: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 15 mg; SAR442168 15 mg/Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.4606, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = -47.38, 95% CI 2-sided [-312.91 to 47.40]
Statistical Analysis 3: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 30 mg; SAR442168 30 mg/Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.9490, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 2.90, 95% CI 2-sided [-138.96 to 60.54]
Statistical Analysis 4: Comparison: Cohort 2: Pooled Placebo vs Cohorts 1 and 2: SAR442168 60 mg; SAR442168 60 mg/Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.2324, Negative binomial regression model; Threshold for significance for p-value was 0.05; Relative reduction in lesions = 65.05, 95% CI 2-sided [-96.21 to 93.77]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs): Weeks 1-4 Period
Description: Adverse event (AE) was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with use of study drug. Serious AE (SAE) was defined as any untoward medical occurrence that, at any dose resulted in death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, disability/incapacity, congenital anomaly/birth defect, or medical event. TEAEs were defined as AEs (serious/non-serious) that developed, worsened, or became serious during on-treatment period (for this outcome measure- "Weeks 1 to 4 period": time from 1st administration of study drug to Week 4). Cohorts 1 and 2 received SAR442168 and placebo for first 4 weeks, respectively.
Time Frame: From Baseline up to Week 4
Population: Analysis was performed on safety population that included all participants from randomized population who had received at least 1 dose or part of dose of study drug. Data was planned to be collected and analyzed on participants at each dose level of SAR442168 in Cohort 1 and pooled population of participants receiving Placebo in Cohort 2 and not planned to be collected during Cohort 1 Placebo administration (Weeks 12 to 16).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: SAR442168 5 mg: Participants who received SAR442168 5 mg orally once daily in Cohort 1.
- Cohort 1: SAR442168 15 mg: Participants who received SAR442168 15 mg orally once daily in Cohort 1.
- Cohort 1: SAR442168 30 mg: Participants who received SAR442168 30 mg orally once daily in Cohort 1.
- Cohort 1: SAR442168 60 mg: Participants who received SAR442168 60 mg orally once daily in Cohort 1.
Arm/Group | Cohort 2: Pooled Placebo | Cohort 1: SAR442168 5 mg | Cohort 1: SAR442168 15 mg | Cohort 1: SAR442168 30 mg | Cohort 1: SAR442168 60 mg
Number analyzed (Participants) | 66 | 16 | 16 | 16 | 16
Participants
  TEAE | 23 | 5 | 3 | 2 | 5
  TESAE | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events: SAR442168 Treatment Period
Description: AE was defined as any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with use of study drug. SAE was defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, persistent disability/incapacity, congenital anomaly/birth defect, or medical event. TEAEs: AEs that developed, worsened, or became serious during on-treatment period (for this outcome measure defined as "SAR442168 treatment period" which was considered as Weeks 1 to 12 for Cohort 1 and Weeks 4 to 16 for Cohort 2).
Time Frame: Weeks 1 to 12 for Cohort 1 participants and Weeks 4 to 16 for Cohort 2 participants
Population: Analysis was performed on safety population. Data was planned to be collected and analyzed on pooled participants at each dose level of SAR442168 (either in Cohort 1 or 2), and was not planned to be collected during placebo administration in either Cohort 1 or 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: SAR442168 5 mg | Cohorts 1 and 2: SAR442168 15 mg | Cohorts 1 and 2: SAR442168 30 mg | Cohorts 1 and 2: SAR442168 60 mg
Number analyzed (Participants) | 33 | 32 | 33 | 32
Participants
  TEAE | 19 | 17 | 18 | 16
  TESAE | 0 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Individual Clinically Relevant Abnormalities in Laboratory Tests (Hematology, Chemistry, Urinalysis), Vital Signs, and Electrocardiograms (ECG)
Description: Individual clinically relevant abnormalities was defined as potentially clinically significant abnormalities (PCSA) considered as SAEs or TEAEs leading to study treatment discontinuation or study discontinuation during the on-treatment period (time from first study drug administration until Week 16), considering all evaluations performed during the on-treatment period that included unscheduled or repeated evaluations.
Time Frame: Baseline up to Week 12 for Cohort 1 participants; Baseline up to Week 4 for Cohort 2 Placebo and from Weeks 4 to 16 for Cohort 2 SAR442168 receiving participants
Population: Analysis was performed on safety population. Data was planned to be collected and analyzed on pooled population of participants at each dose level of SAR442168 (either in Cohort 1 or 2), and pooled population of participants receiving Placebo in Cohort 2 and was not planned to be collected during placebo administration in Cohort 1 (Weeks 12 to 16).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Pooled Placebo | Cohorts 1 and 2: SAR442168 5 mg | Cohorts 1 and 2: SAR442168 15 mg | Cohorts 1 and 2: SAR442168 30 mg | Cohorts 1 and 2: SAR442168 60 mg
Number analyzed (Participants) | 66 | 33 | 32 | 33 | 32
Participants
  Hematology | 0 | 0 | 0 | 0 | 0
  Chemistry | 0 | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0 | 0
  Vitals | 0 | 0 | 0 | 0 | 0
  ECGs | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from the first dose of study drug until the end of the study (Week 16) regardless of seriousness or relationship to study drug
Description: Reported AEs are TEAEs that developed, worsened, or became serious during the treatment-emergent period (time from the first dose of study treatment until the last study visit). Analysis was performed on safety population. Data is reported for pooled populations of Cohort 1 and 2 for each dose of study drug, i.e., events during the 12 weeks of SAR442168 treatment, and for all participants who received placebo either in Cohort 1 or 2 during the placebo treatment period.
Groups:
- Cohort 1 and 2: SAR442168 5 mg: All participants who received SAR442168 5 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohort 1 and 2: SAR442168 15 mg: All participants who received SAR442168 15 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohort 1 and 2: SAR442168 30 mg: All participants who received SAR442168 30 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohort 1 and 2: SAR442168 60 mg: All participants who received SAR442168 60 mg orally once daily for 12 weeks (either in Cohort 1 or 2) during the 16 weeks treatment period.
- Cohort 1: Pooled Placebo: All participants in Cohort 1 who received placebo matching to SAR442168 orally once daily in Weeks 12-16 during the 16 weeks treatment period.
Arm/Group | Cohort 1 and 2: SAR442168 5 mg | Cohort 1 and 2: SAR442168 15 mg | Cohort 1 and 2: SAR442168 30 mg | Cohort 1 and 2: SAR442168 60 mg | Cohort 1: Pooled Placebo | Cohort 2: Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32 | 0/33 | 0/32 | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32 | 0/33 | 1/32 | 0/64 | 0/66
Other Adverse Events (participants affected / at risk) | 19/33 | 17/32 | 18/33 | 16/32 | 10/64 | 23/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 and 2: SAR442168 5 mg (N=33) | Cohort 1 and 2: SAR442168 15 mg (N=32) | Cohort 1 and 2: SAR442168 30 mg (N=33) | Cohort 1 and 2: SAR442168 60 mg (N=32) | Cohort 1: Pooled Placebo (N=64) | Cohort 2: Pooled Placebo (N=66)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 and 2: SAR442168 5 mg (N=33) | Cohort 1 and 2: SAR442168 15 mg (N=32) | Cohort 1 and 2: SAR442168 30 mg (N=33) | Cohort 1 and 2: SAR442168 60 mg (N=32) | Cohort 1: Pooled Placebo (N=64) | Cohort 2: Pooled Placebo (N=66)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy To Animal (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grief Reaction (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 3 (3) | 1 (1) | 4 (7) | 2 (2) | 4 (4)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine Without Aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Muscle Spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix Inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual Headache (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystic Lymphangioma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Fatigue Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Immunoglobulin M Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reticulocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT03889639/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT03889639/SAP_001.pdf